CLINICAL TRIAL: NCT03005262
Title: Expanded Access To MLN8237, For An Individual Patient With Adenocarcinoma Of The Prostate (CTMS# 16-0122)
Brief Title: MLN8237 for a Subject With Adenocarcinoma of the Prostate
Status: No longer available | Type: Expanded Access
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: CTMS 16-0122
Record Dates: First submitted 2016-12-22; First posted 2016-12-29 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — MLN 8237

INTERVENTIONS:
Drug: MLN8237
  Other Names: Alisertib

SUMMARY:
To allow a patient continued access to MLN8237

DETAILED DESCRIPTION:
Expanded access to MLN8237 for an individual patient with adenocarcinoma of the prostate

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Histologically or cytologically confirmed advanced tumors and candidates for docetaxel treatment
* Measurable or evaluable disease is required. Patients must have clinical evidence of progressive disease or persistent disease
* Patients with castration-resistant prostate cancer (CRPC) are required to have
* Pathologically confirmed adenocarcinoma of the prostate
* Evidence of metastatic disease on bone scan or other imaging. Patients with PSA elevation as the only manifestation of disease are not eligible.
* Progressive disease after at least 1 hormonal treatment with documented testosterone levels less than 50 ng/dl
* Concurrent use of an agent for testosterone suppression (e.g., LHRH agonist) is required if the patient has not been surgically castrated
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Recovered to less than or equal to Grade 1 toxicity (CTCAE), to patient's baseline status (except alopecia) or deemed irreversible from the effects of prior cancer therapy and must have evidence of progressive or persistent disease
* Adequate bone marrow, liver and renal function
* Any use of opiates must be stable for at least 2 weeks prior to study entry
* Male patients who agree to practice effective barrier contraception during the entire study and through 6 months after the last dose of study drug OR agree to abstain from heterosexual intercourse
* Voluntary written consent
* Willing to comply with scheduled visits, treatment plan, laboratory tests and other trial procedures
* Suitable venous access for blood sampling

Exclusion Criteria:

* Antineoplastic therapy or any experimental therapy within 21 days before the first dose of MLN8237
* Prior or current investigational therapies within 4 weeks before the first dose of MLN8237
* Radiotherapy to greater than 40% of bone marrow or any radiotherapy (except localized, small field radiation) within 4 weeks prior to enrollment, unless reviewed and approved by the medical monitor
* Nitrosoureas or mitomycin-C within 6 weeks before the first dose of MLN8237.
* Autologous stem cell transplant within 3 months before the first dose of MLN8237, or prior allogeneic stem cell transplant at any time.
* Use of enzyme-inducing antiepileptic drugs such as phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort within 14 days prior to the first dose of MLN8237
* For CRPC patients:
* Radiotherapy or antiandrogen therapy for prostate cancer within 4 weeks prior to enrollment
* Prior treatment with antineoplastic chemotherapy or radioisotopes for advanced prostate cancer
* Use of products known to affect PSA levels within 4 weeks of enrollment
* Major surgery within 4 weeks of study enrollment
* Uncontrolled high blood pressure
* Patients with abnormal gastric or bowel function or who require continuous treatment with antacids or proton pump inhibitors
* Patients receiving chronic steroid therapy other than the following: low dose steroid for the control of nausea and vomiting, topical steroid, inhaled steroid or use of dexamethasone
* Known severe hypersensitivity to docetaxel or other drugs formulated in polysorbate 80
* Comorbid condition or unresolved toxicity that would preclude administration of docetaxel
* Prior history of Grade 2 or greater neurotoxicity or any toxicity that has not resolved to Grade 1 or below
* Symptomatic brain or other CNS metastasis
* Diagnosis or treatment of another malignancy within 2 years preceding first dose of study drug except nonmelanoma skin cancer or in situ malignancy completely resected
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Patients requiring full systemic anticoagulation
* Prior allogeneic bone marrow or other organ transplant
* Active infection requiring systemic therapy within 14 days preceding first dose, or other serious infection
* History of hemorrhagic or thrombotic cerebrovascular event in the past 12 months
* Serious medical or psychiatric illness that could interfere with protocol completion
* Inability to swallow oral medication
* Prior treatment with more than 3 myelosuppressive cytotoxic chemotherapy regimens
* Prior treatment with more than 1 prior taxane-containing regimen

Ages: 18 Years to 100 Years | Sex: Male
Age Groups: Adult, Older Adult